CLINICAL TRIAL: NCT04506450
Title: Peripheral Nerve Block vs Spinal Anesthesia in Hip Surgery: a Randomized Study
Brief Title: Peripheral Nerve Block vs Spinal Anesthesia in Hip Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Università Politecnica delle Marche (Other)
Responsible Party: Principal Investigator, Diego Tavoletti, Principal Investigator, Università Politecnica delle Marche
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 721
Record Dates: First submitted 2020-08-06; First posted 2020-08-10 (Actual); Last update posted 2020-08-10 (Actual); Status verified 2020-08

CONDITIONS: Hip Arthroplasty
Keywords: Regional anesthesia; Hip arthroplasty; Nerve block; Lumbar plexus block
MeSH Terms: interventions — Anesthesia, Spinal

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peripheral nerve block (Active Comparator): The participant will receive a combination of lumbar plexus block, sciatic nerve block, lateral femoral cutaneous nerve block and lateral branch of iliohypogastric nerve block
  Interventions: Procedure: Peripheral nerve block
- Spinal anesthesia (Active Comparator): The participant will receive a combination of spinal anesthesia and lumbar plexus block
  Interventions: Procedure: Spinal anesthesia

INTERVENTIONS:
Procedure: Peripheral nerve block — In this group, four nerve blocks will be associated to ensure adequate anesthesia and analgesia during hip surgery.
  Lumbar plexus and sciatic nerve blocks will be performed with a needle connected to an electrical nerve stimulation. The needle will be advanced until contraction of the femoral quadriceps muscle and plantar or dorsal flexion of the foot will be detected respectively. For both, a mixture of mepivacaine and levobupivacaine will be injected.
  Lateral femoral cutaneous nerve block will be performed with the ultrasound technique. After identifying the nerve, a needle will be inserted with an "in plane" approach and will be injected.
  Lateral branch of iliohypogastric nerve block will be executed with the "De Visme approach". Along the iliac crest (range between 7 and 11 cm from the anterior superior iliac spine) a needle will be inserted until bone contact is found. Then a mixture of mepivacaine and levobupivacaine will be injected.
  Arms: Peripheral nerve block
Procedure: Spinal anesthesia — In this group, spinal anesthesia will be performed to ensure anesthesia during surgery, while lumbar plexus block will be performed to ensure postoperative analgesia Spinal anesthesia will be performed with a 25 G needle and 12 mg 0.5% levobupivacaine will be injected.
  Lumbar plexus block will be performed with a needle connected to an electrical nerve stimulation. The needle will be advanced until contraction of the femoral quadriceps muscle will be detected. 20 ml 0.5% levobupivacaine will be injected.
  Arms: Spinal anesthesia

SUMMARY:
Anesthesia plays an important role in the patient's outcome: each anesthesiological technique has a different cardiovascular impact, because they act differently on the autonomic nervous system, which in turn regulates heart rate, myocardial contractility and vascular tone.

Subarachnoid anesthesia can result in a reduction in cardiac output, hypotension and bradycardia due to blockage of the nerve fibers of the sympathetic system, while peripheral nerve block is associated with a lower impact on the autonomic nervous system, therefore less influence on hemodynamic changes compared to subarachnoid anesthesia.

Hypotension can lead to myocardial ischaemia, especially in patients at high surgical risk.

In addition, peripheral nerve block allows for better coverage from postoperative pain compared to subarachnoid anesthesia in patients undergoing hip surgery.

This leads to less postoperative stress, with less impact on cardiac and respiratory function.

Numerous studies have shown the efficacy and safety of regional anesthesia in hip surgery.

This study aims to compare the hemodynamic changes of subarachnoid anesthesia and peripheral nerve block in patients who underwent total and partial hip replacement

DETAILED DESCRIPTION:
All patients who meet the inclusion and exclusion criteria will be enrolled. Enrolled patients will be informed of the study modality. In case of a favorable opinion, the patient will be made to sign the informed consent. Subsequently a code will be assigned to the patient for randomization.

There are two randomization groups: in the PNB group the patient will undergo lumbar plexus block, sciatic nerve block, lateral femoral cutaneous nerve block and lateral branch of iliohypogastric nerve block, while in the SA group, the patient will undergo subarachnoid anesthesia and lumbar plexus block.

In the preoperative room, ECG, pulseoximetry will be estabilished and an arterial radial cannula will be inserted under local anesthesia to monitor blood pressure. A premedication with midazolam (0.05-0.1 mg / kg) will be administered before anesthesia is performed.

At this point, the type of anesthesia will be followed on the basis of the randomization group.

The following variables will be evaluated:

* hemodynamic parameters in the perioperative period
* onset time of the sensory and motor block
* fluids and vasoactive drugs administered
* anesthesiological complications
* degree of patient satisfaction
* duration of surgery
* degree of postoperative pain and analgesic therapy administered
* mini mental state evaluation (in the preoperative and postoperative period)
* start physical rehabilitation
* clinical complications during hospitalization
* duration of hospitalization

ELIGIBILITY:
Inclusion Criteria:

* Subject has signed and dated an Informed Consent Form
* Subject is classified as a ASA (American Society of Anesthesiologists) status I-IV
* Subject is age 18- 99 years old
* Patients undergoing total hip arthroplasty

Exclusion Criteria:

* Subject inability to provide adequate informed consent
* Study refusal
* Age younger than 18 years
* Contraindication to regional anesthesia
* Allergy to local anesthetics
* Neurological disease of the lower limbs
* Moderate or severe dementia disease
* Psychiatric disease

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Change of the systolic blood pressure | During anesthetic and surgery procedures
  Systolic blood pressure will be evalueted after sedation, at the end of the anesthestic procedure, and then every 2.5 minutes up to the 20th minute. Then at the beginning of the surgery and every 5 minutes until the end of the surgery
Change of the diastolic blood pressure | During anesthetic and surgery procedures
  Diastolic blood pressure will be evalueted after sedation, at the end of the anesthestic procedure, and then every 2.5 minutes up to the 20th minute. Then at the beginning of the surgery and every 5 minutes until the end of the surgery
Change of the mean blood pressure | During anesthetic and surgery procedures
  Mean blood pressure will be evalueted after sedation, at the end of the anesthestic procedure, and then every 2.5 minutes up to the 20th minute. Then at the beginning of the surgery and every 5 minutes until the end of the surgery
Change of the heart rate | During anesthetic and surgery procedures
  Heart rate will be evalueted after sedation, at the end of the anesthestic procedure, and then every 2.5 minutes up to the 20th minute. Then at the beginning of the surgery and every 5 minutes until the end of the surgery

SECONDARY OUTCOMES:
Change in the onset time of the nerve block | Up to 20 minutes
  Sensitivity to the lower limbs will be assessed by pinprick test and cold test after the end of the anesthetic procedure
Change in the degree of the sensory block | Up to 20 minutes after the end of the anesthetic procedure
  Sensitivity to the lower limbs will be assessed by pinprick test and cold test after the end of the anesthetic procedure
Change of the Motor block degree | Up to 20 minutes after the end of the anesthetic procedure
  The motor block will be assessed by the Bromage scale after the end of the anesthetic procedure. Grade 1: complete block (unable to move feet or knees). Grade 2: almost complete block (able to move feet only). Grade 3: partial block (just able to move knees). Grade 4: detectable weakness of hip flexion (between score 3 and 5). Grade 5: No detectable weakness of hip flexion while supine (full flexion of knees). Grade 6: able to perform partial knee bend.
Amount ephedrine administered during the perioperative period | During anesthetic and surgery procedures
  Ephedrine use, mg.
Amount atrophine administered during the perioperative period | During anesthetic and surgery procedures
  Atropine use, mg.
Amount Fluids administered during the perioperative period | During anesthetic and surgery procedures
  All fluids administered, ml.
Degree of patient satisfaction | At the end of surgery
  the degree of patient satisfaction will be measured on a scale ranging from 0 to 3 (0= bad; 1= not bad; 2=good; 3=excellent)
Duration of surgery | During surgery
  minutes
Postoperative pain score | 1, 3, 6, 12, 24, 36, 48 hours after the end of surgery
  11-point numeric rating scale ranging from '0' representing one extreme (e.g. "extremely dissatisfied") to '10' representing the other extreme (e.g. "extremely satisfied")
Amount of analgesic drugs administered | 1, 3, 6, 12, 24, 36, 48 hours after the end of surgery
  Paracetamol use, mg; Morphine use, mg; Ketorolac use, mg.
Assessment of mental state | Preoperative; 24 hours after the end of surgery; 48 h after the end of surgery, 72 h after the end of surgery and 96 h after the end of surgery.
  It will be evaluated through the mini mental state evaluation
Beginning of physical rehabilitation | Immediately after the surgery
  number of day
Anesthetic and surgery complications | During anesthetic and surgery procedures
  Assessment for existence of complications related to procedures in form of Y/N (such as hypotension, bradycardia, local anesthetic epidural spread, local anesthetic systemic toxicity, nausea and vomiting
Clinical complications | Immediately after the surgery
  Assessment for existence of complications related to procedures in form of Y/N (such as neuropathy, nausea and vomiting, heart and vascular diseases, respiratory dysfunction, urinary retention, renal failure, cognitive disorder, death
Duration of hospitalization | Up to one month
  Duration (day) of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Diego Tavoletti, MD, Principal Investigator — Ospedali riuniti di Ancona-Università politecnica delle Marche
Locations (1):
- Ospedali Riuniti di Ancona - Università politecnica delle marche, Ancona, Italy